CLINICAL TRIAL: NCT00871130
Title: The Effect of Bariatric Surgery on Thyroid Function and Morphology, a Retrospective Study
Brief Title: The Effect of Bariatric Surgery on Thyroid Function and Morphology
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Vanessa Banz, MD, Department of Visceral and Transplant Surgery, Bern University Hospital
Other Study IDs: KEK_13_01_09
Record Dates: First submitted 2009-03-24; First posted 2009-03-30 (Estimated); Last update posted 2009-03-30 (Estimated); Status verified 2009-03

CONDITIONS: Thyroid Function; Obesity
Keywords: Thyroid gland; bariatric surgery; weight loss; thyroid hormones; adult; morbid obesity; cohort
MeSH Terms: conditions — Obesity; Thyroid Diseases; Weight Loss; Obesity, Morbid | interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Bariatric surgery — gastric banding, gastric bypass or vertical gastroplasty either open or laparoscopic or a combination of any

SUMMARY:
The aim is to evaluate the effect of dramatic weight loss after bariatric surgery on thyroid function (thyroid hormone levels and particulary morphological changes) in the short and long-term setting of a cross-sectional study. A particular focus will be made with regard to putting into correlation preoperative thyroid function abnormalities and postoperative changes over time with respect to the type of bariatric intervention carried out.

DETAILED DESCRIPTION:
Background:

Over the last decades, there has been an increase in obesity in virtually all population groups with approximately 1.6 billion adults worldwide estimated to be overweight in 2005 and 400 million of these people qualifying as being obese.

Although hormonal disturbances may play a certain role in the development of obesity, more important are the possible consequences of obesity and the influence of surgically-induced rapid weight loss on overall endocrine function of these patients. Studies evaluating the effect of weight loss on thyroid function show inconsistent results. Whilst some authors have shown that weight loss after bariatric surgery may have a positive effect on thyroid dysfunction, especially in individuals with preoperative subclinical hypothyroidism 1 resulting in normalisation of TSH levels, others fail to show any significant postoperative changes.

Objective:

To evaluate the effect of dramatic weight loss after bariatric surgery on thyroid function (thyroid hormone levels and particularly morphological changes) in the short and long-term in the setting of a cross-sectional study. A particular focus will be made with regard to putting into correlation preoperative thyroid function abnormalities and postoperative changes over time with respect to the type of bariatric intervention carried out.

Methods:

BMI, thyroid hormones (TSH, fT3, fT4 levels), need for thyroxin substitution (or equivalent medication) as well as pre- and postoperative morphological changes in the thyroid gland (usually via sonography)and Leptin values will be assessed retrospectively.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent bariatric surgery between 1998 and 2007

Exclusion Criteria

* age >18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who have received a surgical procedure to result in desired weight reduction (gastric banding, gastric bypass or vertical gastroplasty either open or laparoscopic or a combination of any)
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 1998-01; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
thyroid hormone levels (change in) | preoperative, 3, 6 and 12 months postoperative

SECONDARY OUTCOMES:
morphological changes of the thyroid gland | up to 12 months postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Banz, MD, Principal Investigator — Dep.of Visceral and Transplant Surgery, Bern University Hospital
Locations (1):
- Dep.of Visceral and Transplant Surgery, Bern University Hospital, Bern, Switzerland

REFERENCES:
- [Background] Chikunguwo S, Brethauer S, Nirujogi V, Pitt T, Udomsawaengsup S, Chand B, Schauer P. Influence of obesity and surgical weight loss on thyroid hormone levels. Surg Obes Relat Dis. 2007 Nov-Dec;3(6):631-5; discussion 635-6. doi: 10.1016/j.soard.2007.07.011. PMID 18023816
- [Background] Alagna S, Cossu ML, Masala A, Atzeni MM, Ruggiu M, Satta FM, Fais E, Rovasio PP, Noya G. Evaluation of serum leptin levels and thyroid function in morbidly obese patients treated with bariatric surgery. Eat Weight Disord. 2003 Jun;8(2):95-9. doi: 10.1007/BF03324997. PMID 12880185
- [Background] Reinehr T, Andler W. Thyroid hormones before and after weight loss in obesity. Arch Dis Child. 2002 Oct;87(4):320-3. doi: 10.1136/adc.87.4.320. PMID 12244007